CLINICAL TRIAL: NCT04632017
Title: Computerized Cardiotocography Monitoring in Fetuses With Preterm Premature Rupture of Membranes
Brief Title: Computerized Cardiotocography Monitoring of Fetuses With pPROM
Acronym: COCA-PROM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Maddalena Morlando, Assistant Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 8452
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cardiotocography; Premature Rupture of Membrane; Rupture of Membranes; Premature; Sepsis; Premature Birth
Keywords: cardiotocography; Premature Rupture of Membrane; computerized cardiotocography; premature birth
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Sepsis; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pPROM: Singleton pregnancies admitted for pPROM to the Obstetrics ward
  Interventions: Diagnostic Test: Computerized cardiotocography
- Control group: Healthy pregnant women matched for gestational age
  Interventions: Diagnostic Test: Computerized cardiotocography

INTERVENTIONS:
Diagnostic Test: Computerized cardiotocography — To compare Dawes and Redman indices as determined by computer analysis of the fetal heart tracing

SUMMARY:
Preterm premature rupture of membranes (PPROM) is associated with neonatal complications leading to a high rate of cerebral palsy, sepsis, and death. Choosing the best time of delivery is crucial to improve fetal outcome. The balance is between a premature delivery exposing the infant to all the risk of prematurity, and keeping the baby in utero, prolonging the exposure to an adverse intrauterine milieu. There are no objective and reproducible tools to help in this decision-making process. Techniques most frequently used for fetal surveillance are biased by high inter- and intra-observer variability. Computerized cardiotocography (cCTG) identifies several objective parameters related to fetal heart rate (FHR) to determine fetal well-being. cCTG has been successfully used in fetuses with intrauterine growth restriction, but it has never been used in prospective studies to assess its role in the management of fetuses with PPROM. The investigators designed a case control study to highlight cCTG differences in PPROM pregnancies versus physiological pregnancies, to establish the effectiveness in predicting adverse outcome, and to develop a score to predict neonatal outcome.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) occurs in 2 to 3% of pregnancies and is associated with higher maternal and neonatal morbidity and mortality. Neonatal complications are primarily due to prematurity and to ascending infection of the amniotic cavity (chorioamnionitis), leading to a high rate of cerebral palsy, intracranial hemorrhage, sepsis, pneumonia, and death. Every physician is confronted with an extremely difficult and at the same time of paramount importance decision, when it comes to establish the timing of the delivery of a premature fetus with PPROM. The balance is between delivering a premature infant exposed to all the risk of prematurity, and keeping the baby in utero, prolonging the exposure to an adverse intrauterine milieu. At present, there are no objective and reproducible tools to help in this decision-making process. The technique most frequently used for fetal surveillance is cardiotocography (CTG). Assessment of the fetal heart rate is classified subjectively as 'reassuring' or 'not reassuring'. Dawes and Redman have suggested computerized CTG (cCTG), which eliminates inter- and intra-observer variability, identifying several objective parameters to determine fetal well-being. After the multicentre TRUFFLE-Study, cCTG became the best tool to manage fetuses with intrauterine growth restriction (IUGR). However, the use of cCTG has never been investigated in prospective studies to assess its role in the management of fetuses with PPROM. Of note, amniotic fluid concentration of glucose, lactate, interleukin-6 (IL-6), and matrix metalloproteinase-8 (MMP-8) have been associated with neonatal septicemia, chorioamnionitis, preterm birth, and/or fetal inflammatory response syndrome in women with pPROM.

ELIGIBILITY:
Inclusion Criteria:

* pPROM between 24 and 34 weeks (w)

Exclusion Criteria:

* multiple pregnancy, structural fetal anomalies, preexisting or gestational diabetes mellitus and\or hypertension, intrauterine growth restriction.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton pregnancies admitted for pPROM to the Obstetrics ward of this Hospital will be recruited after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Preterm birth rate | Less than 37 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
Preterm birth rates | Less than 24, 28, 34 weeks gestation
Birth weight | Time of delivery
  Weight of the baby at the time of delivery
Low birth weight rate | Time of delivery
  Birth weight <2500g
Neonatal death rate | Between birth and 28 days of age
Composite adverse neonatal outcomes | Between birth and 28 days of age
  Number of neonates who will have at least one of the following:
  necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH) (grade 3 or higher), respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), retinopathy (ROP), blood-culture proven sepsis and neonatal death
Maternal outcomes | Between birth and 28 days after the birth
  Number of mothers who will have at least one of the following:
  sepsis, histological chorioamnionitis, hysterectomy, intensive care unit admission.
Dawes and Redman indices | between 24 and 34 weeks of gestation
  determined by computer analysis of the fetal heart tracing

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Schiattarella, MD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided